CLINICAL TRIAL: NCT03425032
Title: Low-dose Whole Body Computed Tomography Scanning
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 16-5477
Record Dates: First submitted 2018-01-31; First posted 2018-02-07 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Computed Tomography; Image Quality
MeSH Terms: interventions — Tomography Scanners, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CT scanner — Regular CT imaging of the abdomen and pelvis
  Other Names: Genesis TSX-350A CT scanner

SUMMARY:
Computed tomography represents the mainstay for diagnosing various diseases in the whole body. Over the past decade, enormous efforts were undertaken by both CT manufacturers and radiologist to reduce the radiation dose to patients. Today, the dose is significantly lower that it was before the era of multislice CT and iterative reconstruction methods. The X-ray beam originating from the tube in a CT system contains a spectrum of different energies, whereby the "harder" beams with higher energy penetrate the patient better, and the "softer" beams will be absorbed through the patient's tissues. Recent research has been shown that the radiation dose can be further reduced by improved primary beam filtering in CT. This study is intended to compare the radiation dose in clinically indicated, routine CT examination while maintaining a diagnostic image quality, on a new CT system with modified primary beam filtering.

DETAILED DESCRIPTION:
At the Joint Department of Medical Imaging (JDMI), the investigators periodically adjust the radiation dose and modify the clinical imaging protocols in order to continuously optimize image quality in CT. The investigators have formalized the process of radiation dose adjustments by implementing a CT dose committee that meets on a monthly basis and reviews imaging protocols (SOP). The committee includes radiologists, technologists, vendor representative (if needed), managers and the radiation protection officer. Part of the review is the investigator's in-house developed Coral image quality review program as well as the clinically used radiation dose monitoring software (Radiometric).

Part of the evaluation study of the new CT system is to monitor 520 patients who will undergo a clinically indicated CT scan on the new system. Identical to standard-of-care (SOC) quality insurance, the investigators will use the existing monitoring software (Radiometric, JDMI) in order to capture the data in the existing database. The investigators will also capture quality data through the existing CT image quality feedback tool. After installation of the new CT system, the investigators will maintain the radiation dose as currently applied in the standard JDMI wide imaging protocols and examine 20 patients on the new system; radiation dose and image quality feedback will be recorded in the identical fashion to standard operating procedures (CT image quality and radiation dose committee). Subsequently, the investigators will drop the dose by approx. 10% for each scanning protocol and scan the subsequent 250 patients while concurrently analyzing the impact on the collective dose to the patient population. Based on the expected increase in image noise, the investigators will calculate the possible additional dose reduction in percent and modify all protocols accordingly for the subsequent 250 patients. This step-down approach ensures that no CT scan will be performed with too little dose, and that all CT scans remain diagnostic.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are clinically scheduled for a CT of the body (any part, or a combination of different parts).

Exclusion Criteria:

* There are no exclusion criteria for the purpose of this study. Patients must able to consent to the study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be routed to the new CT system in sequential order and as per clinical schedule. There will be no specific inclusion criteria for the study.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Radiation dose | Through study completion, an average of 1 year
  Mean radiation dose (DLP), comparison to existing data (Radimetrics database)

CONTACTS AND LOCATIONS:
Overall Officials: Patrik Rogalla, Principal Investigator — UHN

IPD SHARING:
Plan to Share IPD: No
Image quality data will be stored in our clinical data base identical to SOC. We will not create a new database for the purpose of the study. Radiation dose measurements will also be stored in our clinical database identical to SOC. The selection of the patients for the purpose of the study (radiation dose to the population) is being performed through the Radimetrics software that sorts the database based on the CT equipment used. We will get a full list of all patients who were scanned on the new system, with a graphical display of the radiation dose distribution in relation to the other clinical CT. This feature is routinely used for all other clinical CT scanner

REFERENCES:
- [Result] Zhang G, Marshall N, Jacobs R, Liu Q, Bosmans H. Bowtie filtration for dedicated cone beam CT of the head and neck: a simulation study. Br J Radiol. 2013 Aug;86(1028):20130002. doi: 10.1259/bjr.20130002. Epub 2013 May 31. PMID 23728948
- [Result] Mail N, Moseley DJ, Siewerdsen JH, Jaffray DA. The influence of bowtie filtration on cone-beam CT image quality. Med Phys. 2009 Jan;36(1):22-32. doi: 10.1118/1.3017470. PMID 19235370
- [Result] Tkaczyk JE, Du Y, Walter D, Wu X, Li J, Toth T. Simulation of CT dose and contrast-to-noise as function of bowtie shape. Proc SPIE 2004;5368:403-410